CLINICAL TRIAL: NCT01558960
Title: Intravitreal Injections of Melphalan for Retinoblastoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sufficient findings to draw conclusions
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RB-001-HMO-CTIL
Record Dates: First submitted 2012-03-01; First posted 2012-03-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2012-03

CONDITIONS: Retinoblastoma
Keywords: Retinoblastoma
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IVit Treatment group (Experimental): Intravitreal injections of Melphalan
  Interventions: Drug: IVit Melphalan

INTERVENTIONS:
Drug: IVit Melphalan — IVit injections of Melphalan

SUMMARY:
Retinoblastoma treatment has become more and more focused in the last years. New treatments developed by Dr. Kaneko from Japan in 1995 are now being tested in clinical trials.

Intra-arterial chemotherapy with Melphalan has shown success in some patients but with limited response when there is marked vitreal seeding. For these cases Intravitreal injections of Melphalan have been successful in Japan.

In this study the same chemotherapy (melphalan) will be administered intravitreally (directly through the eye wall) and the response (short and long term) will be monitored.

DETAILED DESCRIPTION:
Intravitreal injections of Melphalan will be given to cases unresponsive to chemotherapy or with vitreal seeding of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Retinoblastoma that has not responded to chemotherapy
* Retinoblastoma that has vitreal seeding

Exclusion Criteria:

* previous failure of IVit Melphalan

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
treatment response | 1 year
  short term response to treatment and long term complications

SECONDARY OUTCOMES:
complications | 1 year
  short and long term complications

CONTACTS AND LOCATIONS:
Overall Officials: Shahar Frenkel, MD, PhD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah-Hebrew University Medical Center, Jerusalem, Israel